CLINICAL TRIAL: NCT06851754
Title: Hormone Replacement Therapy in Adolescents With Premature Ovarian Insufficiency
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10002141; 002141-CH
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Premature Ovarian Insufficiency
Keywords: Premature Ovarian Insufficiency; Hormone Replacement Therapy; Adolescents; Bone Health
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Progesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (No Intervention): Healthy Control Participants
- POI Patients (Experimental): POI patients will be receiving transdermal 17 beta-estradiol and oral micronized progesterone.
  Interventions: Drug: Progesterone; Drug: Estrogen Patch

INTERVENTIONS:
Drug: Progesterone — Oral micronized progesterone will be added (100 mg/day for 12 days/month) in the event of spontaneous vaginal bleeding and/or at 12 months over the 2-year protocol.
  Arms: POI Patients
Drug: Estrogen Patch — participants with POI (n=85) will receive transdermal 17 beta-estradiol (beginning at a dose of 25 microgram/patch applied weekly), with the dose increased at 3 months to 50 microgram, and thereafter every 6 months to 75 and 100 microgram/patch for pubertal induction or estrogen replacement (with 100 microgram/patch representing a full adolescent or young adult estradiol dose). The continued escalation of the estradiol dose and patch strength will be guided by the clinical presentation and physical examination (by the PI or designated AI).
  Arms: POI Patients

SUMMARY:
Background:

Premature ovarian insufficiency (POI) is a condition in which women under the age of 40 years have absent or irregular menstrual cycles. POI can cause infertility, signs of menopause, osteoporosis, and other symptoms. Hormone replacement therapy (HRT) is a treatment that gives women extra hormones, such as estrogen and progesterone. HRT works well in adult women. Researchers want to find the most effective doses and regimens for adolescents.

Objective:

To monitor the effects of HRT on adolescents with POI.

Eligibility:

Female adolescents aged 11 to 19 years diagnosed with POI. Healthy volunteers are also needed.

Design:

All participants will have clinic visits every 6 months for 2 years. Each visit may last 2 days. Each visit may include:

Blood and urine tests.

A test of their heart function.

A test to measure the stiffness of their blood vessels. Participants will lie flat with a blood pressure cuff on a leg and a meter on the neck while the cuff inflates.

A test of their grip strength. Participants will squeeze a handheld device as hard as they can.

Two scans to measure bone density. For one, participants will lie on a table while a scanner passes along their body. For the other, participants will sit in a chair and insert their forearm, then their lower leg, into a scanner.

A test to measure skin pigmentation. Participants skin will be touched lightly with a device.

An optional visual exam of the vagina. Some vaginal fluid may also be collected with a cotton swab/cytobrush.

Participants with POI will receive HRT. They will be given estrogen patches and progesterone pills.

DETAILED DESCRIPTION:
Study Description:

This is a study of adolescents with premature ovarian insufficiency (POI) and their response to hormone replacement therapy (HRT).

Objectives:

Primary:

To identify the phenotype and associated genotype of adolescents with POI at the time of diagnosis, including assessment of overall bone health of participants pre- and post-HRT treatment with respect to bone mineral density (BMD) and other skeletal endpoints.

Bone Health:

-Follow patients with POI for bone health assessments:

* Measure BMD at different skeletal sites, including the central skeleton (lumbar spine, total body less head, and hip - femoral neck and total hip)
* Perform vertebral fracture assessment (VFA)
* Determine body composition of lean body and fat mass (total body) and correlate with BMD.
* Assess skin pigmentation and muscle grip strength and correlate with BMD

Secondary:

Bone Health

-Follow patients with POI for bone health assessments:

* Measure BMD at peripheral skeleton (radius and tibia)
* Evaluate bone microarchitecture and strength of the radius and tibia.

Metabolic Phenotype:

* Follow patients with POI for metabolic assessment:

  * Insulin resistance
  * Cardiovascular risk
  * Lipid profiles
  * Bone turnover

Muscle Phenotype:

-Follow patients with POI for muscle function assessment:

* Determine hand grip muscle strength
* Evaluate lean body mass (by DXA) to determine muscle mass

Cardiovascular Health

-Follow patients with POI for a cardiovascular evaluation:

* Electrophysiologic parameters (from 12-lead EKG)
* Arterial stiffness (by Pulse Wave Velocity, PWV)
* Coagulation studies to determine the impact of HRT on clotting function

Genetic profiling:

-If obtained, assess the baseline genotype of patients with POI to correlate with BMD and other health outcomes

--If subjects are co-enrolled on NIAID protocol 17I0122, utilize that genetic sequencing data to associate with genotype and response of multiple health outcomes to HRT.

Quality of Life:

-Follow patients with POI for evaluation of an individual s perception of their life quality and health:

* Evaluate the individual s perceived occupational performance in self-care, productivity, and leisure
* Evaluate the individual s occupations or hobbies that align with their interests

Psychological health:

-Follow patients with POI for evaluation of an individual s mood and well-being:

* Measure symptoms and severity of depression
* Measure the state and trait components of anxiety

Menopause profile:

-Follow patients with POI for determining signs and symptoms of menopause:

* Evaluate reproductive hormonal changes
* Assess menopausal symptoms and their severity
* Evaluate vaginal health

Hormone Replacement Therapy:

-Follow patients with POI longitudinally to determine the most effective HRT management:

* Evaluate dosage, delivery, combination of HRT
* Evaluate effects of HRT on bone, cardiovascular, metabolic, gynecologic, and psychological health

Endpoints:

Primary:

Longitudinal evaluation of BMD of the central skeleton (lumbar spine).

As secondary measures of bone health, dual-energy x-ray absorptiometry (DXA) measures of skeletal sites other than the spine (DXA - hip/total body) will be evaluated longitudinally in POI participants and their BMD compared to healthy control participants. Using DXA, vertebral fractures assessment (VFA) will be performed in POI participants and compared to healthy control participants. In addition, BMD will be evaluated with respect to skin pigmentation and muscle grip strength.

Secondary:

* High-resolution peripheral quantitative computed tomography (HRpQCT) bone density and strength measures by HRpQCT of the peripheral skeleton (radius and tibia) will be evaluated longitudinally in participants with POI and their BMD compared to healthy control participants.
* Compare metabolic and cardiovascular parameters in participants with POI to healthy controls.
* Compare muscle phenotype in participants with POI to healthy controls by measuring muscle strength using hand grip dynamometry and measuring lean body mass (as measure of total body muscle mass) by DXA.
* Compare repolarization changes (by 12-lead EKG), arterial stiffness (by PWV) and coagulation parameters in participants with POI to healthy controls.
* Compare genetic background of participants with POI to healthy controls using whole genome sequencing.
* Evaluate quality of life with Canadian Occupational Performance Measure (COPM) and Interest Checklist questionnaires.
* Evaluate psychological health of participants with POI compared to healthy controls using the Beck Depression Inventory and Spielberger State/Trait Anxiety Inventory.
* Evaluate menopausal profile in participants with POI compared to healthy controls by detecting changes in ovarian hormonal levels and correlating with responses on the Menopause Rating Scale, and vaginal cytology and degree of atrophy after HRT compared to baseline (and participants vs. controls).
* Compare health effects from a typical clinical HRT regiment over the course of 2 years of administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for POI Participants

To be eligible to participate in this study, an individual must meet all the following criteria:

* Individuals aged 11-19 years, inclusive, at the time of enrollment.
* Diagnosis of premature ovarian insufficiency.
* Documentation of two elevated serum FSH measurements, at least month apart, greater than the testing laboratory s the upper reference range (for age/Tanner stage).
* Identify as female (i.e., sex assigned at birth)
* Negative pregnancy test.

Inclusion Criteria for Healthy Volunteers:

* Individuals aged 11-19 years.
* Identify as female (i.e., sex assigned at birth)
* Negative pregnancy test.
* Absence of known chronic disease

EXCLUSION CRITERIA:

Male participants are excluded from both study groups (POI and Healthy Volunteers) as POI affects only the female reproductive system, while pregnant participants are not eligible to have DXA or HRpQCT imaging for safety reasons.

Exclusion Criteria for POI participants:

An individual who meets any of the following criteria will be excluded from participation in this study:

* POI in the setting of Turner syndrome.
* Patients who screened positive for celiac disease.
* Receipt of any medications including HRT determined by the investigator to affect bone metabolism 3 months prior to enrollment.
* Any medical condition determined by the investigator to affect bone health will be excluded.
* Presence of a medical, psychiatric, or social condition which, in the opinion of the investigator, would place undue burden on the subject, NIH resources, or increase risk of participation.
* Report of sexual activity but refusal to use a copper intrauterine device or double barrier forms of contraception during the study.

Exclusion Criteria for Healthy Volunteers:

For healthy volunteers, all exclusion criteria will apply as for POI participants except for number 1.

Ages: 11 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 185 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2031-12-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal evaluation of BMD of the central skeleton (lumbar spine). | 2 years
  measures of bone health, dual-energy x-ray absorptiometry (DXA) measures of skeletal sites other than the spine (DXA - hip/total body) will be evaluated longitudinally in POI participants and their BMD compared to healthy control participants. Using DXA, vertebral fractures assessment (VFA) will be performed in POI participants and compared to healthy control participants. In addition, BMD will be evaluated with respect to skin pigmentation and muscle grip strength.

SECONDARY OUTCOMES:
Evaluate bone density and strength of the radius and tibia in participants with POI and compare with healthy controls. | 2 years
  Bone Health - Evaluate bone density and strength of the radius and tibia in participants with POI and compare with healthy controls.
Compare metabolic and cardiovascular parameters between participants with POI and healthy controls. | 2 years
  Metabolic Phenotype - Compare metabolic and cardiovascular parameters between participants with POI and healthy controls.
Assess muscle strength and lean body mass in participants with POI compared to healthy controls. | 2 years
  Muscle Phenotype - Assess muscle strength and lean body mass in participants with POI compared to healthy controls.
Analyze heart repolarization, arterial stiffness, and coagulation parameters in participants with POI versus healthy controls. | 2 years
  Cardiovascular Health - Analyze heart repolarization, arterial stiffness, and coagulation parameters in participants with POI versus healthy controls.
Compare the genetic background of participants with POI to healthy controls using whole genome sequencing. | 2 years
  Genetic profiling - Compare the genetic background of participants with POI to healthy controls using whole genome sequencing.
Assess quality of life using COPM and Interest Checklist questionnaires. | 2 years
  Quality of Life - Assess quality of life using COPM and Interest Checklist questionnaires.
Evaluate psychological health using the Beck Depression Inventory and Spielberger State/Trait Anxiety Inventory. | 2 years
  Psychological Health - Evaluate psychological health using the Beck Depression Inventory and Spielberger State/Trait Anxiety Inventory.
Compare menopausal profile, including ovarian hormone levels and responses to the Menopause Rating Scale, between participants with POI and healthy controls. | 2 years
  Menopausal profile - Compare menopausal profile, including ovarian hormone levels and responses to the Menopause Rating Scale, between participants with POI and healthy controls.
Assess health effects of a typical clinical HRT regimen over two years. | 2 years
  Hormone Replacement Therapy - Assess health effects of a typical clinical HRT regimen over two years.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Gordon, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be deposited into a data repository in line with NIH regulations.
Supporting Information: SAP, Analytic Code
Time Frame: In line with publication of results.
Access Criteria: De-identified datasets used to generate results presented in manuscripts will be deposited into a repository that can be publicly accessible in line with NIH regulations. In compliance with ethical standards and institutional policies, other access to individual participant data will be governed by a structured data-sharing framework to ensure participant privacy and confidentiality. Access to IPD will be granted under a Data Use Agreement that specifies permissible uses, prohibits re-identification or further data sharing, and requires secure storage and handling of data. Access will be restricted to de-identified or coded datasets, with direct identifiers removed.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002141-CH.html